CLINICAL TRIAL: NCT02520349
Title: Lab to Real World Assessment of E-cigarette Abuse Liability and Appeal
Status: Completed | Type: Observational
Sponsor: Truth Initiative (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Jennifer Pearson, Research Investigator, Truth Initiative
Other Study IDs: 5K01DA037950 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma nicotine: Investigators will examine change in plasma nicotine concentration before and after 5 minutes of directed product use (10 total puffs). At the start of the session, a phlebotomist will draw 7mL of blood via venipuncture (no catheter). Participants will then be directed to take a puff of their own brand/assigned e-cigarette device every 30 seconds for 5 minutes. At the end of the directed use session, the phlebotomist will draw another 7mL of blood via venipuncture. Blood samples will be processed at the Center for Study of Tobacco Products lab, frozen, and walked across the street to the Bioanalytical Mass Spectrometry Core Laboratory at VCU for cotinine/3-OH analysis using previously developed assays. Blood samples will not be retained for additional analyses.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MarkTen and e-Go e-cigarettes

SUMMARY:
The proposed research is a longitudinal human lab study to examine how measures of abuse liability and product appeal vary by e-cigarette device type, and how these lab assessments may predict subsequent e-cigarette and other tobacco use behavior at 1,3, and 6 months. An additional aim is to evaluate e-cigarette safety and tolerability among smokers by device type.

DETAILED DESCRIPTION:
The proposed research is a longitudinal human lab study to involving 6 lab visits and 3 follow-up surveys at 1, 3, and 6 months after participants' last lab visit. Investigators will enroll 30 smokers (≥10 cig/day) who have not used e-cigarettes in the past 30 days and have never used e-cigarettes "fairly regularly." After a telephone screening to confirm eligibility, participants will attend Virginia Commonwealth University's (VCU) Clinical Behavioral Pharmacology Laboratory for all lab visits. The specific aims are to:

Aim 1. Examine how measures of abuse liability and product appeal vary by ECIG device type (Markten vs. e-Go).

Aim 2. Compare differences in abuse liability and product appeal between participants' usual brand of tobacco cigarette, Markten, and e-Go.

Aim 3. As an exploratory aim, examine the extent to which measures of abuse liability and product appeal as measured in the lab (including TPPT) predict participants' real-world ECIG use at the 1-, 3-, and 6-month follow-up surveys.

Aim 4. To monitor safety and tolerability the MarkTen and e-Go among smokers.

ELIGIBILITY:
Inclusion Criteria:

1. be between 18-65 years of age;
2. reside in the Richmond metro area;
3. be proficient in English;
4. be interested in trying e-cigarettes, assessed at the initial screening;
5. have no immediate plans (in the next 30 days) to quit smoking;
6. have an active email address (for online follow-up surveys);
7. report current cigarette use (≥10 CPD for ≥1 year). To biochemically confirm cigarette smoking status, eligible participants must have an exhaled carbon monoxide (CO) of ≥15ppm at screening using a Vitalograph CO monitor.

Exclusion Criteria:

Individuals fitting any of the following criteria will not be eligible to participate.

1. Individuals who have used e-cigarettes in the past 30 days;
2. Individuals who used e-cigarettes more than 5 times in their lives;
3. Individuals with uncontrolled or unstable medical or psychiatric conditions;
4. Individuals with current or recent (within 6 months) drug/alcohol abuse;
5. Individuals who weigh less than 110 lbs;
6. Individuals with conditions that would require medical attention during the course of the study (such as hypertension [systolic BP over 140, diastolic BP over 90] or elevated heart rate [over 90 BPM]);
7. Women who are currently pregnant/breastfeeding or who have plans to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 30 community volunteers who currently use 10 or more cigarettes per day and have no immediate plans to quit smoking will be enrolled. Investigators will attempt to recruit an equal number of men and women of diverse racial/ethnic backgrounds. This preliminary study is not intended to address gender or race/ethnic differences.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in blood nicotine concentration | 3 weeks - before and after product administration
  A phlebotomist will draw 7mL of blood via venipuncture (no catheter) before and after directed tobacco product use at Lab Visits 2-6.
Nicotine withdrawal symptom alleviation | 3 weeks - before and after product administration
  Participants will answer questions about their nicotine withdrawal symptoms (e.g. headache, tired, etc)
Change in subjective tobacco product appeal | 3 weeks - before and after product administration
  Participants will answer questions about the positive and negative physical effects of using the product and how much they like the product.
Change in heart rate | 3 weeks - before and after product administration
  Participants' heart rate (HR) will be monitored continuously during Lab Visits 2-6. Participants will commence physiological data measurement 30 minutes before the start of the directed tobacco use bout to establish a resting HR.
Number of Participants with Adverse Events by ECIG Device Type as a Measure of Safety and Tolerability | 3 weeks - before and after product administration
  A count of the number of participants who report adverse events associated with the study, such as headache, chest pain, cough/sputum, nausea/vomiting, dizziness, confusion/stupor, feeling sick, sore throat, shortness of breath, abdominal pain, pleurisy, blurry vision, and tiredness, by e-cigarette device type.
Change in blood pressure | 3 weeks - before and after product administration
  Participants' blood pressure (BP) will be monitored continuously during Lab Visits 2-6. Participants will commence physiological data measurement 30 minutes before the start of the directed tobacco use bout to establish resting BP.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Pearson, PhD, Principal Investigator — Truth Initiative
Locations (2):
- United States (2):
  - American Legacy Foundation, Washington D.C., District of Columbia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes